CLINICAL TRIAL: NCT02751086
Title: Prospective, Observational, Multicenter Study on Minimally Invasive Gastrectomy for Gastric Cancer: Robotic, Laparoscopic and Open Surgery Compared on Operative and Follow-up Outcomes
Brief Title: Robotic, Laparoscopic and Open Gastrectomy Compared on Short and Long Term Outcomes
Acronym: IMIGASTRICII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Study Group on Minimally Invasive Surgery for Gastric Cancer (Other)
Responsible Party: Principal Investigator, Amilcare Parisi, Principal Investigator, International Study Group on Minimally Invasive Surgery for Gastric Cancer
Other Study IDs: 002
Record Dates: First submitted 2016-04-10; First posted 2016-04-26 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer
Keywords: minimally invasive surgery; gastrectomy; robotic surgery; laparoscopic surgery; laparoscopy; robot-assisted; robotic; robotic gastrectomy; laparoscopic gastrectomy; minimally invasive gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Robotic Gastrectomy: Patients who will be treated for gastric cancer with the assistance of the robotic surgical system
  Interventions: Procedure: Robotic Gastrectomy
- Laparoscopic Gastrectomy: Patients who will be treated for gastric cancer through laparoscopic devices.
  Interventions: Procedure: Laparoscopic Gastrectomy
- Open Gastrectomy: Patients who will be treated for gastric cancer with traditional open surgery.

INTERVENTIONS:
Procedure: Robotic Gastrectomy — Minimally invasive surgical approach, related to the availability of a robotic surgical system (eg Da Vinci surgical system), that allows a surgeon to perform surgery through a console and dedicated devices.
  Groups: Robotic Gastrectomy
Procedure: Laparoscopic Gastrectomy — Minimally invasive surgical approach performed through traditional laparoscopy.
  Groups: Laparoscopic Gastrectomy

SUMMARY:
The overall purpose is to develop and maintain a multi-institutional database comprising of information regarding surgical, clinical and oncological features of patients that will be treated for gastric cancer with robotic, laparoscopic or open approaches and subsequent follow-up.

The main objective is to compare the three surgical arms on surgical and clinical outcomes, as well as on the oncological follow-up.

DETAILED DESCRIPTION:
A review of the scientific literature, which was recently published by the IMIGASTRIC study group, aimed to perform a more complete analysis of the current situation regarding performing minimally invasive surgery for gastric cancer. Significant limitations were found in the analyzed studies, including:

* Small samples of patients, mostly low-quality comparative studies
* Selection bias in the comparison groups (e.g. stage, extent of lymphadenectomy)
* Absence of subgroup analysis in significant research fields
* Lack of information on the surgical techniques adopted

A large prospective multicenter registry could thus be the optimal way to clarify the role of minimally invasive surgery for gastric cancer and permit the evaluation of its short and long-term effects. A working basis for analyzing outcomes of interest and obtaining directions for guidelines and future study developments can also be created. The following would be the main advantages of a large prospective multicenter registry:

* Achieving a large sample of patients
* Collecting multiple variables, allowing for the making of a comprehensive statistical report
* Standardizing the methodology to be adopted, thus increasing accuracy
* Bringing together the experiences of both East and West to discover shared points A prospective registry can become a powerful tool that can guide research in this field to new developments and pave the way for other investigational opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric cancer
* Preoperative staging work-up performed by upper endoscopy and/or endoscopic ultrasound, and CT scan and in accordance to international guidelines
* Early Gastric Cancer
* Advanced Gastric Cancer
* Patients treated with curative intent in accordance to international guidelines

Exclusion Criteria:

* Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, Krukenberg tumors, involvement of other organs
* Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score > 4
* History of previous abdominal surgery for gastric cancer
* Synchronous malignancy in other organs
* Palliative surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with gastric cancer eligible for curative surgery.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with intraoperative adverse events | During surgery
  events other than the normal course of the surgery
Mean of retrieved lymph nodes | Within 30 days after surgery
  Count of retrieved lymph nodes at the histopathological examination of the surgical specimen
Rate of patients alive | 1 year after surgery
  subjects alive at the planned endpoint
Rate of patients alive | 2 year after surgery
  subjects alive at the planned endpoint
Rate of patients alive | 3 year after surgery
  subjects alive at the planned endpoint
Rate of patients alive | 4 year after surgery
  subjects alive at the planned endpoint
Rate of patients alive | 5 year after surgery
  subjects alive at the planned endpoint

SECONDARY OUTCOMES:
Mean post-operative hospital stay | from the day after surgery to patient discharge, assessed up to 90 days
  hospital stay of the patients after surgery
Rate of complications after discharge | 5 year after surgery
  any surgical related event after patient's discharge

CONTACTS AND LOCATIONS:
Overall Officials: Amilcare Parisi, MD, Principal Investigator — St. Mary's Hospital of Terni
Locations (1):
- Department of Digestive Surgery, St. Mary's Hospital, University of Perugia, Terni, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parisi A, Nguyen NT, Reim D, Zhang S, Jiang ZW, Brower ST, Azagra JS, Facy O, Alimoglu O, Jackson PG, Tsujimoto H, Kurokawa Y, Zang L, Coburn NG, Yu PW, Zhang B, Qi F, Coratti A, Annecchiarico M, Novotny A, Goergen M, Lequeu JB, Eren T, Leblebici M, Al-Refaie W, Takiguchi S, Ma J, Zhao YL, Liu T, Desiderio J. Current status of minimally invasive surgery for gastric cancer: A literature review to highlight studies limits. Int J Surg. 2015 May;17:34-40. doi: 10.1016/j.ijsu.2015.02.021. Epub 2015 Mar 7. PMID 25758348
- [Background] Parisi A, Desiderio J. Establishing a multi-institutional registry to compare the outcomes of robotic, laparoscopic, and open surgery for gastric cancer. Surgery. 2015 Apr;157(4):830-1. doi: 10.1016/j.surg.2014.12.007. Epub 2015 Jan 26. No abstract available. PMID 25633739
- [Background] Desiderio J, Jiang ZW, Nguyen NT, Zhang S, Reim D, Alimoglu O, Azagra JS, Yu PW, Coburn NG, Qi F, Jackson PG, Zang L, Brower ST, Kurokawa Y, Facy O, Tsujimoto H, Coratti A, Annecchiarico M, Bazzocchi F, Avanzolini A, Gagniere J, Pezet D, Cianchi F, Badii B, Novotny A, Eren T, Leblebici M, Goergen M, Zhang B, Zhao YL, Liu T, Al-Refaie W, Ma J, Takiguchi S, Lequeu JB, Trastulli S, Parisi A. Robotic, laparoscopic and open surgery for gastric cancer compared on surgical, clinical and oncological outcomes: a multi-institutional chart review. A study protocol of the International study group on Minimally Invasive surgery for GASTRIc Cancer-IMIGASTRIC. BMJ Open. 2015 Oct 19;5(10):e008198. doi: 10.1136/bmjopen-2015-008198. PMID 26482769
- [Background] Marano A, Choi YY, Hyung WJ, Kim YM, Kim J, Noh SH. Robotic versus Laparoscopic versus Open Gastrectomy: A Meta-Analysis. J Gastric Cancer. 2013 Sep;13(3):136-48. doi: 10.5230/jgc.2013.13.3.136. Epub 2013 Sep 30. PMID 24156033
- [Background] Vinuela EF, Gonen M, Brennan MF, Coit DG, Strong VE. Laparoscopic versus open distal gastrectomy for gastric cancer: a meta-analysis of randomized controlled trials and high-quality nonrandomized studies. Ann Surg. 2012 Mar;255(3):446-56. doi: 10.1097/SLA.0b013e31824682f4. PMID 22330034
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2010 (ver. 3). Gastric Cancer. 2011 Jun;14(2):113-23. doi: 10.1007/s10120-011-0042-4. No abstract available. PMID 21573742
- [Background] Japanese Gastric Cancer Association. Japanese classification of gastric carcinoma: 3rd English edition. Gastric Cancer. 2011 Jun;14(2):101-12. doi: 10.1007/s10120-011-0041-5. No abstract available. PMID 21573743
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Waddell T, Verheij M, Allum W, Cunningham D, Cervantes A, Arnold D. Gastric cancer: ESMO-ESSO-ESTRO clinical practice guidelines for diagnosis, treatment and follow-up. Eur J Surg Oncol. 2014 May;40(5):584-591. doi: 10.1016/j.ejso.2013.09.020. No abstract available. PMID 24685156
- [Background] Washington K. 7th edition of the AJCC cancer staging manual: stomach. Ann Surg Oncol. 2010 Dec;17(12):3077-9. doi: 10.1245/s10434-010-1362-z. No abstract available. PMID 20882416
- See also: Study's website. The study is open to other interested Institutions. — http://www.imigastric.com
- Available data/document: Study Protocol, study information, news — http://www.imigastric.com — The study is open to other interested Institutions. Correspondance to: Jacopo Desiderio, MD djdesi85@hotmail.it